CLINICAL TRIAL: NCT02131415
Title: Canadian Non-Interventional Prospective Cohort Study on the Real - Life Assessment of Abilify Maintena ™ in Schizophrenia
Brief Title: Real Life Assessment of Abilify Maintena
Acronym: ReLiAM
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment combined with positive preliminary results
Sponsor: Lundbeck Canada Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15914N
Record Dates: First submitted 2014-04-11; First posted 2014-05-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; real-life; long-acting injectable; Reliam
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional, Canadian, study in patients treated with Abilify Maintena™ for schizophrenia followed for 24 months, with 9 visits recommended. Study assessments and administration of questionnaires will take place during the patient regular assessments or injection visits that are part of routine care. The main objective of the study is to describe the impact of treatment with Abilify Maintena™ on global functional status.

DETAILED DESCRIPTION:
* Treatment

  * All patients will be treated with Abilify Maintena™ administered once monthly at the dose that is as per the treating physician's judgment.
  * The assignment of the patients to be treated with Abilify Maintena™ is not decided in advance by the study protocol and is clearly separated from the decision to include the patients in the study. For all patients that will be included in the study, the decision to initiate treatment with Abilify Maintena™ must have been reached prior to and independently of enrolling the patient in the study.
  * Any treatment is to be prescribed according to the recommendations given in the approved Canadian Product Monograph.
* Study Sites

  - Up to 30 sites planned in Canada: Patients will be recruited by community or hospital based psychiatrists. A random representative sample of Canadian psychiatrists will be identified as the sampled population of physicians that will be invited to participate in the study and will undergo a feasibility assessment. Those that satisfy the feasibility assessment, have adequate volume of patients and are willing to participate in the study will be enrolled.
* Data Collection and Handling

  - All patient data will be collected by the site investigator or designated staff and will be entered in an electronic data capture (EDC) system that will be developed for the study. Patient questionnaires will be completed during the visit using paper-based surveys. The questionnaire data will be transcribed into the study database by the CRO personnel using a double data entry system. There will be no patient identifying information recorded in any of the study data collection forms or databases. All patients will be identified using encrypted random study ID numbers. Data monitoring and source verification will be conducted on a sample of patients. Auditing of patient qualification will also be conducted on a sample of patients within each site.
* Missing data handling

  - There will be no imputation for missing data. General linear models with repeated measures and mixed effects will be used to compensate for unequal follow up intervals and missing data points. All analyses will be conducted on observed cases.
* Safety analyses - The safety population will comprise all patients included in the study that have had at least one treatment with Abilify Maintena™. Adverse events will be described with the MedDRA dictionary of terms classified by preferred term and system - organ class.

ELIGIBILITY:
Inclusion Criteria

* The patient must be 18 (19 for patients from British Columbia) years of age or older.
* The patient must have been diagnosed with schizophrenia.
* The patient must be at least mildly ill (CGI-S score of ≥3).
* The treating physician must have reached the decision to treat the patient with Abilify Maintena™ prior to and independently of soliciting the patient to participate in the study.
* The patient and legal guardian (if applicable and when allowable by law) must have signed an informed consent indicating the understanding of the study and allowing the use of their anonymous data for the purposes of the study.
* The patient and caregiver(s) (if applicable) must be fluent in English or French, in order to be able to complete the questionnaires.

Exclusion Criteria

* The patient does not comprehend or refuses to sign the informed consent.
* The patient has any contraindications to the use of Abilify Maintena™ as specified in the Canadian Product Monograph.
* The patient has previously received one or more doses of Abilify Maintena™.
* The patient presents a significant suicidal risk as judged by the investigator.
* The patient is a pregnant or lactating female.
* The patient is a member of the study personnel or of their immediate families, or is a subordinate (or immediate family member of a subordinate) to any of the study personnel.
* The patient has previously been enrolled in this study.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with Abilify Maintena™ for schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
The change in GAF score while on treatment with Abilify Maintena™ for 12 months | from baseline to 12 months

SECONDARY OUTCOMES:
The change in score on CGI-I and CGI-S at various timepoints over 24 months. | from baseline to 3, 6, 9, 12,15,18, 21,24 months
The change in GAF score at various time points over 24 months | from baseline to 3, 6, 9,15, 18, 21, 24 months.
Number of patients achieving remission, amount of time it takes to achieve remission, amount of time they remain in remission and the rates of relapse. | from baseline to 3, 6, 9,12,15,18, 21, 24 months
Number of injections of Abilify Maintena™ received over the course of 24 months, in order to describe adherence | at 3, 6, 9,12,15,18, 21, 24 months
Number of patients with Adverse Events as a measure of safety and tolerability. | At 3, 6, 9,12,15,18, 21, 24 months
The change in SOFAS score while on treatment with Abilify Maintena™. | from baseline to 3, 6 ,9 ,12 ,15 ,18 ,21 ,24 months

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (17):
- Canada (17):
  - CA012, Calgary, Alberta
  - CA008, Penticton, British Columbia
  - CA017, Vancouver, British Columbia
  - CA006, Halifax, Nova Scotia
  - CA011, Brockville, Ontario
  - CA001, Chatham, Ontario
  - CA014, Kingston, Ontario
  - CA004, Kitchener, Ontario
  - CA013, London, Ontario
  - CA016, Mississauga, Ontario
  - CA010, Ottawa, Ontario
  - CA002, Windsor, Ontario
  - CA009, Montreal, Quebec
  - CA003, Montreal, Quebec
  - CA015, Montreal, Quebec
  - CA005, Québec, Quebec
  - CA019, Rivière-du-Loup, Quebec

REFERENCES:
- [Derived] Roy MA, Therrien F, Boucher M, Oluboka O. Long-term effectiveness of aripiprazole once monthly on functioning and quality of life in schizophrenia: results of year 2 of the ReLiAM study. BMC Psychiatry. 2024 Nov 14;24(1):797. doi: 10.1186/s12888-024-06240-x. PMID 39538234
- [Derived] Oluboka O, Clerzius G, Janetzky W, Schottle D, Therrien F, Wiedemann K, Roy MA. Improvement of functioning in patients with schizophrenia: real-world effectiveness of aripiprazole once-monthly (REACT study). BMC Psychiatry. 2023 May 31;23(1):383. doi: 10.1186/s12888-023-04893-8. PMID 37259053
- [Derived] Schottle D, Janetzky W, Therrien F, Wiedemann K. BPRS domains, items and subgroups analyses, and CGI-I ratings in pooled data from non-interventional studies of aripiprazole once-monthly in schizophrenia (REACT study). BMC Psychiatry. 2023 Mar 14;23(1):162. doi: 10.1186/s12888-023-04651-w. PMID 36918846
- [Derived] Margolese HC, Boucher M, Therrien F, Clerzius G. Treatment with aripiprazole once-monthly injectable formulation is effective in improving symptoms and global functioning in schizophrenia with and without comorbid substance use - a post hoc analysis of the ReLiAM study. BMC Psychiatry. 2022 Dec 8;22(1):773. doi: 10.1186/s12888-022-04397-x. PMID 36482352
- [Derived] Schottle D, Clerzius G, Janetzky W, Oluboka O, Roy MA, Therrien F, Wiedemann K. Real-world effectiveness of aripiprazole once-monthly REACT study: Pooled analysis of two noninterventional studies. Eur Psychiatry. 2022 Jul 20;65(1):e42. doi: 10.1192/j.eurpsy.2022.27. PMID 35855645
- [Derived] Mustafa S, Bougie J, Miguelez M, Clerzius G, Rampakakis E, Proulx J, Malla A. Real-life assessment of aripiprazole monthly (Abilify Maintena) in schizophrenia: a Canadian naturalistic non-interventional prospective cohort study. BMC Psychiatry. 2019 Apr 16;19(1):114. doi: 10.1186/s12888-019-2103-x. PMID 30991969